CLINICAL TRIAL: NCT00946101
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of MEDI3414 in Children
Brief Title: A Study to Evaluate the Safety of HIN1 Monovalent Vaccine (MEDI3414) in Children 2 to 17 Years of Age
Acronym: MI-CP217
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Elissa Malkin, D.O., MedImmune LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP217; HHS/ASPR (Other Grant/Funding Number: HHSO100200900002I)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: randomized, double-blind, placebo-controlled
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDI3414 [Influenza A (H1N1) vaccine] (Active Comparator): MEDI3414- Monovalent vaccine was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 FFU (fluorescent focus units) of influenza virus type A/California/07/2009.
  Interventions: Biological: MEDI3414 [Influenza A(H1N1) live attenuated, intranasal]
- Placebo (Placebo Comparator): Placebo - Placebo was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI3414 [Influenza A(H1N1) live attenuated, intranasal] — 0.5 mL: (intranasal sprayer)
  Arms: MEDI3414 [Influenza A (H1N1) vaccine]
Biological: Placebo — Placebo was supplied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the safety and descriptive immunogenicity of the H1N1 influenza vaccine in healthy children.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety and descriptive immunogenicity of a monovalent influenza virus vaccine containing a new 6:2 influenza virus reassortant in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2 to 17 years of age (not yet reached their 18th birthday) at the time of randomization
* Healthy by medical history and physical exam
* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU and written informed assent) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Females of child-bearing potential, (ie, unless premenarchal, surgically sterile [eg, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy], has sterile male partner, or practices abstinence) must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of investigational product, and must agree to continue using such precautions for 60 days after the second dose of investigational product. In addition, the subject must also have a negative urine or blood pregnancy test at screening and, if screening and Day 1 do not occur on the same day, on the day of vaccination prior to randomization. Investigator judgment is required to assess the childbearing potential of a pre-adolescent or adolescent girl.
* Males, unless not sexually active, must use an effective method of birth control with a female partner and must agree to continue using such contraceptive precautions for at least 30 days after the second dose of investigational product (from Day 1 through Day 59 of the study)
* Subject's legal representative available by telephone
* Subject/subject's legal representative is able to understand and comply with the requirements of the protocol, as judged by the investigator
* Ability to complete follow-up period of 180 days after Dose 2 as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of the investigational product including egg or egg protein, gelatin or arginine, or serious, life-threatening, or severe reactions to previous influenza vaccinations
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (> 100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
* History of asthma, or in children < 5 years of age, history of recurrent wheezing
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* A household contact who is severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); subject should additionally avoid close contact with severely immunocompromised individuals for at least 21 days after receipt of investigational product
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after the second dose of investigational product (use of licensed agents for indications not listed in the package insert is permitted)
* Use of aspirin or salicylate-containing products within 30 days prior to randomization or expected receipt through 30 days after final vaccination
* Expected receipt of antipyretic or analgesic medication (non-salicylate-containing) on a daily or every other day basis from randomization through 14 days after receipt of each dose of investigational product
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after administration of each dose of investigational product
* Receipt of any nonstudy vaccine within 30 days before or after Dose 1 or expected receipt of any nonstudy vaccine within 30 days before or after Dose 2
* Known or suspected mitochondrial encephalomyopathy
* Adolescent subject is pregnant or a nursing mother
* Any condition (eg, chronic cough, allergic rhinitis) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Subject, legal representative, or immediate family member of subject is an employee of the clinical study site or is otherwise in involved with the conduct of the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Malkin, D.O., Study Director — MedImmune LLC
Locations (16):
- United States (16):
  - Coastal Clinic Research, Inc., Mobile, Alabama
  - Benchmark Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - Benchmark Research, San Francisco, California
  - Kentucky Pediatric Research Center, Bardstown, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Rochester Clinical Research Inc., Rochester, New York
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Benchmark Research, Austin, Texas
  - Benchmark Research Ft. Worth, Fort Worth, Texas
  - Benchmark Research San Angelo, San Angelo, Texas

REFERENCES:
- [Derived] Mallory RM, Malkin E, Ambrose CS, Bellamy T, Shi L, Yi T, Jones T, Kemble G, Dubovsky F. Safety and immunogenicity following administration of a live, attenuated monovalent 2009 H1N1 influenza vaccine to children and adults in two randomized controlled trials. PLoS One. 2010 Oct 29;5(10):e13755. doi: 10.1371/journal.pone.0013755. PMID 21060780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participation began once written informed consent was obtained. The first and last dates of informed consent were 03 Aug 2009 and 19 Aug 2009. Once informed consent was obtained, a subject identification number was assigned using an interactive voice response system, and screening evaluations began to assess study eligibility.
Pre-assignment Details: Eligible subjects were randomly assigned in a 4:1 ratio to receive 2 doses of study monovalent vaccine or placebo by intranasal spray; the doses were administered approximately 28 days apart, on Days 1 and 29.
Groups:
- H1N1 Monovalent Influenza Vaccine: MEDI3414- Monovalent vaccine supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units (FFU) of influenza virus type A/California/07/2009. Subjects were to receive two doses by intranasal spray; each dose was administered approximately 28 days apart on Days 1 and 29.
- Placebo: Placebo - 0.5 mL of sucrose-phosphate buffer contained in intranasal sprayers. Subjects were to receive a total of 2 doses by intranasal spray; each dose was administered approximately 28 days apart on Days 1 and 29.
Period: Overall Study
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Started | 261 (Intent to Treat population, enrolled and randomized) | 65
Day 15 Post Dose 1 | 260 | 64
Day 15 Post Dose 2 | 254 | 63
Completed | 257 | 63
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal of consent | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 261 | 65 | 326
Age Continuous [Mean (Standard Deviation); unit: years] | 8.9 (4.3) | 9.2 (4.3) | 9.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 36 | 166
  Male | 131 | 29 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 17 | 67
  Not Hispanic or Latino | 211 | 48 | 259
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 43 | 12 | 55
  White | 198 | 43 | 241
  More than one race | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
  Other | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fever Post Dose 1 (Days 1-8), Defined as an Axillary Temperature ≥ 101°F (38.3°C).
Description: The number of participants with fever between the two treatment groups was compared based on the upper limit of the two-sided 95% exact confidence intervals for the rate difference (Vaccine minus Placebo). The upper limit of the two-sided 95% confidence intervals was evaluated against the prespecified equivalence criterion of 10% which corresponded to the following hypotheses: H0 (null): rate difference ≥ 10%, HA (alternative): rate difference < 10%.
Time Frame: Days 1- 8
Population: The safety population included all participants who received at least one dose of investigational product and experienced any follow-up for safety (H1N1=259; Placebo=65).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 4 | 1
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; The rate of subjects with fever between the two treatment groups was compared based on the upper limit of the two-sided 95% exact confidence intervals for the rate difference (Vaccine minus Placebo). The upper limit of the two-sided 95% confidence intervals was evaluated against the pre-specified equivalence criterion of 10% which corresponds to the following hypotheses: H0 (null): rate difference ≥ 10%, HA (alternative): rate difference < 10%; Test type: Non-Inferiority or Equivalence — For the calculation of the power to rule out a 10% increase of fever rate in vaccine recipients with 300 evaluable subjects (240 vaccine and 60 placebo recipients), it is assumed that the true fever rate in the monovalent vaccine group is 3.0% to 8.0%,and the true fever rate in placebo group is 0% to 3% lower than the fever rate in the vaccine group; score; rate difference = 0.0, 95% CI 2-sided [-6.4 to 3.1]

2. Primary Outcome: Number of Participants Who Experience a Post Dose 1 (Day 15) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: Seroresponse is described as greater than or equal to a 4-fold rise in hemagglutination inhibition (HAI) titer from baseline. All immunogenicity analyses was based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: Participants who received Dose 1 of study vaccine (H1N1=259; Placebo=65), had valid HAI measurements from blood samples obtained at baseline and post Dose 1 were included in the analysis (H1N1=129; Placebo=32).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 129 | 32
participants | 10 | 2
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; The number of subjects who experienced a post-dose seroresponse was compared based on the upper limit of the two-sided 95% exact confidence intervals for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 1.5, 95% CI 2-sided [-12.8 to 9.8]

3. Primary Outcome: Number of Participants Who Experience a Post Dose 1 (Day 29) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: Seroresponse is described as greater than or equal to a 4-fold rise in HAI titer from baseline. All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: Participants who received Dose 1 of study vaccine (H1N1=259; Placebo=65) and had valid HAI measurements from blood samples obtained at baseline and post Dose 1 (H1N1=126; Placebo=32).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 126 | 32
participants | 14 | 2
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; score; rate difference = 4.9, 95% CI 2-sided [-9.6 to 13.8]

4. Primary Outcome: Number of Participants Who Experience a Post Dose 2 (Day 57) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: as for outcome 3
Time Frame: Day 1, Day 57
Population: Participants who received 2 doses of the same study vaccine (H1N1=258; Placebo=65) and had valid HAI measurements from blood samples obtained at baseline and post Dose 2 were included in the analysis (H1N1=250; Placebo=62).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 250 | 62
participants | 80 | 9
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; score; rate difference = 17.5, 95% CI 2-sided [5.5 to 27.1]

5. Secondary Outcome: Number of Participants With Any Solicited Symptoms Within 7 Days After Vaccination With Investigational Product, Dose 1
Description: Other solicited symptoms include fever (> 100°F [37.8°C] axillary), runny/stuffy nose, sore throat, cough, headache, generalized muscle aches, decreased activity level (lethargy) or tiredness/weakness, decreased appetite.
Time Frame: Days 1-8
Population: The safety population included all participants who received at least one dose of investigational product (H1N1=259; Placebo=65), experienced any follow-up for safety and had solicited symptoms data available during the reporting period (H1N1=259; Placebo=65).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 97 | 21
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; Rates of solicited symptoms following each dose (Days 1 to 8 and Days 1 to 15) between the two treatment groups were compated following each dose. Exact two-sided 95% confidence intervals (Chan and Zhang, 1999) on the rate difference (Vaccine minus Placebo) were constructed. There were no prespecified equivalence criteria for the secondary analyses; Test type: Superiority or Other; score; rate difference = 5.1, 95% CI 2-sided [-8.4 to 17.6]

6. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs) Within 7 Days After Vaccination With Investigational Product, Dose 1
Time Frame: Days 1-8
Population: The safety population included all participants who received at least one dose of investigational product (H1N1=259; Placebo=65) and experienced any follow-up for safety (H1N1=259; Placebo=65).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 28 | 7

7. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 7 Days After Vaccination With Investigational Product, Dose 1
Time Frame: Days 1-8
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 18 | 1

8. Secondary Outcome: Number of Participants With Any Solicited Symptoms Within 14 Days After Vaccination With Investigational Product, Dose 1
Time Frame: Days 1-15
Population: The safety population included all participants who received at least one dose of investigational product (H1N1=259; Placebo=65), experienced any follow-up for safety, and had solicited symptoms data available during the reporting period (H1N1=259; Placebo=65).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 122 | 22
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; Rates of solicited symptoms following each dose (Days 1 to 8 and Days 1 to 15) between the two treatment groups were compared following each dose. Exact two-sided 95% confidence intervals (Chan and Zhang, 1999) on the rate difference (Vaccine minus Placebo) were constructed. There were no prespecified equivalence criteria for the secondary analyses; Test type: Superiority or Other; score; rate difference = 13.3, 95% CI 2-sided [-0.4 to 25.7]

9. Secondary Outcome: Number of Participants Reporting AEs Within 14 Days After Vaccination With Investigational Product, Dose 1
Time Frame: Days 1-15
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 47 | 11

10. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 14 Days After Vaccination With Investigational Product, Dose 1
Time Frame: Days 1-15
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 27 | 2

11. Secondary Outcome: Number of Participants With Any Solicited Symptoms Within 7 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-36
Population: The safety population for solicited symptoms Dose 2 included all participants who received Dose 2 (H1N1=258; Placebo=65), experienced any follow-up for safety and had solicited symptom data available during the reporting period (H1N1=255; Placebo=63).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 65 | 20
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; score; rate difference = -6.3, 95% CI 2-sided [-19.7 to 6.1]

12. Secondary Outcome: Number of Participants Reporting AEs Within 7 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-36
Population: The safety population included all participants who received Dose 2 (H1N1=258; Placebo) and experienced any follow-up for safety (H1N1=255; Placebo=63).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 20 | 2

13. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 7 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-36
Population: The safety population included all participants who received Dose 2 (H1N1=258; Placebo=65) and experienced any follow-up for safety (H1N1=255; Placebo=63).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 10 | 5

14. Secondary Outcome: Number of Participants With Any Solicited Symptoms Within 14 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-43
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 93 | 27
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; score; rate difference = -6.4, 95% CI 2-sided [-20.3 to 7.1]

15. Secondary Outcome: Number of Participants Reporting AEs Within 14 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-43
Population: The safety population included all participants who received Dose 2 (H1N1=258; Placebo=65), experienced any follow-up for safety (H1N1=255; Placebo=63).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 35 | 9

16. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 14 Days After Vaccination With Investigational Product, Dose 2
Time Frame: Days 29-43
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 22 | 11

17. Secondary Outcome: Number of Participants With New Onset Chronic Diseases (NOCDs) Within 28 Days After Vaccination With Investigational Product, Dose 1.
Description: An NOCD was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant. Examples of NOCDs included, but were not limited to, diabetes, asthma, autoimmune disease (eg, lupus, rheumatoid arthritis), and neurological disease (eg, epilepsy, autism). Examples of events not considered NOCDs were mild eczema, diagnosis of a congenital anomaly present at study entry, or acute illness (eg, otitis media, bronchitis).
Time Frame: Days 1-29
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 0 | 0

18. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Within 28 Days After Vaccination With Investigational Product, Dose 1
Description: SAEs were those AEs that resulted in death; were immediately life threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly in the offspring of a participant; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization and that, based on appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Days 1-29
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 1 | 0

19. Secondary Outcome: Number of Participants With NOCDs Within 28 Days After Vaccination With Investigational Product, Dose 2.
Description: as for outcome 17
Time Frame: Days 29-57
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 0 | 1

20. Secondary Outcome: Number of Participants With SAEs Within 28 Days After Vaccination With Investigational Product, Dose 2
Description: as for outcome 18
Time Frame: Days 29-57
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 255 | 63
participants | 0 | 0

21. Secondary Outcome: Number of Participants With NOCDs Within 180 Days Post Final Dose of Investigational Product.
Description: as for outcome 17
Time Frame: Days 1-209
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
Participants | 0 | 1

22. Secondary Outcome: Number of Participants With SAEs Within 180 Days Post Final Dose of Investigational Product.
Description: as for outcome 18
Time Frame: Days 1-209
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 65
participants | 2 | 1

23. Secondary Outcome: Number of Participants Who Achieve a Post Dose 1 (Day 15) HAI Titer Greater Than or Equal to 32 Against the H1N1 Strain in All Participants, Regardless of Baseline Serostatus.
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 129 | 32
participants | 13 | 1
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine; The number of subjects who achieved a post Dose 1 HAI titer greater than or equal to 32 against the H1N1 strain was compared based on the upper limit of the two-sided 95% exact confidence intervals for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 7.0, 95% CI 2-sided [-6.1 to 14.7]

24. Secondary Outcome: Number of Participants Who Achieve a Post Dose 1 (Day 29) HAI Titer Greater Than or Equal to 32 Against the H1N1 Strain in All Participants, Regardless of Baseline Serostatus.
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: Participants who received Dose 1 of study vaccine (H1N1=259; Placebo=65), had valid HAI measurements from blood samples obtained at baseline and post Dose 1 were included in the analysis (H1N1=126; Placebo=32).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 126 | 32
participants | 13 | 1
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; score; rate difference = 7.2, 95% CI 2-sided [-5.8 to 15.1]

25. Secondary Outcome: Number of Participants Who Achieve a Post Dose 2 (Day 57) HAI Titer Greater Than or Equal to 32 Against the H1N1 Strain in All Participants, Regardless of Baseline Serostatus.
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 57
Population: Participants who received 2 doses of the same study vaccine (H1N1=258; Placebo=65), had valid HAI measurements from blood samples obtained at baseline and post Dose 2 were included in the analysis (H1N1=250; Placebo=62).
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 250 | 62
participants | 66 | 6
Statistical Analysis 1: Comparison: H1N1 Monovalent Influenza Vaccine vs Placebo; The number of subjects who achieved a post Dose 2 HAI titer greater than or equal to 32 against the H1N1 strain was compared based on the upper limit of the two-sided 95% exact confidence intervals for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 16.7, 95% CI 2-sided [5.9 to 25.2]

26. Secondary Outcome: Serum HAI Geometric Mean Titers (GMTs) in All Participants, Regardless of Baseline Serostatus, Dose 1 (Day 15)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 129 | 32
titer | 3.55 [2 to 128] | 2.89 [2 to 32]

27. Secondary Outcome: Serum HAI GMTs in All Participants, Regardless of Baseline Serostatus, Dose 1 (Day 29)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: as for outcome 24
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 126 | 32
titer | 3.53 [2 to 512] | 2.71 [2 to 64]

28. Secondary Outcome: Serum HAI GMTs in All Participants, Regardless of Baseline Serostatus, Dose 2 (Day 57)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 57
Population: as for outcome 25
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | H1N1 Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 250 | 62
titer | 7.61 [2 to 4096] | 3.70 [2 to 128]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 14 days after each vaccination, ie, Days 1-15 and Days 29-43. Serious adverse events (SAEs) were collected through 28 days after each vaccination, ie, Days 1-28 and Days 29-57 and through 180 days post last dose.
Description: Telephone contacts were made by site personnel to the participant/participant's parent or legal guardian at various times during the study to assess safety.
Groups:
- H1N1 Monovalent Vaccine Days 1-28; H1N1 Monvalent Vaccine Days 29-57; H1N1 Monovalent Vaccine Days 58-209: MEDI3414- Monovalent vaccine supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units (FFU) of influenza virus type A/California/07/2009.
- Placebo Days 1-28; Placebo Days 29-57; Placebo Days 58-209: Placebo - 0.5 mL of sucrose-phosphate buffer contained in intranasal sprayers
Arm/Group | H1N1 Monovalent Vaccine Days 1-28 | Placebo Days 1-28 | H1N1 Monvalent Vaccine Days 29-57 | Placebo Days 29-57 | H1N1 Monovalent Vaccine Days 58-209 | Placebo Days 58-209
Serious Adverse Events (participants affected / at risk) | 1/259 | 0/65 | 0/255 | 0/63 | 1/259 | 1/65
Other Adverse Events (participants affected / at risk) | 13/259 | 2/65 | 11/255 | 3/63 | 0/255 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | H1N1 Monovalent Vaccine Days 1-28 (N=259) | Placebo Days 1-28 (N=65) | H1N1 Monvalent Vaccine Days 29-57 (N=255) | Placebo Days 29-57 (N=63) | H1N1 Monovalent Vaccine Days 58-209 (N=259) | Placebo Days 58-209 (N=65)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/255 (0) | 0/63 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/255 (0) | 1/63 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/255 (1) | 0/63 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Monovalent Vaccine Days 1-28 (N=259) | Placebo Days 1-28 (N=65) | H1N1 Monvalent Vaccine Days 29-57 (N=255) | Placebo Days 29-57 (N=63) | H1N1 Monovalent Vaccine Days 58-209 (N=255) | Placebo Days 58-209 (N=63)
nausea (Gastrointestinal disorders) | 5 (6) | 2 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.